CLINICAL TRIAL: NCT06310668
Title: Has CBT an Effect on Emotional Intelligence in Patients With Substance Use Disorder?: A Randomized Clinical Trial
Brief Title: Has CBT an Effect on Emotional Intelligence in Patients With Substance Use Disorder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Medical Syndicate (Other)
Responsible Party: Principal Investigator, Hassan Mohammed Sonbol, lecturer of psychiatry (principal investigator), Egyptian Medical Syndicate
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT IN substance use disorder
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT intervention arm (Experimental): patients with substance use disorder in the inpatient department of the addiction unit in Mansoura University Hospital who will receive group CBT sessions
  Interventions: Behavioral: group cognitive behavioral therapy sessions
- NON-CBT control arm (No Intervention): age and gender-matched patients with substance use disorder in the outpatient clinics of the addiction unit in Mansoura University Hospital who will not receive group CBT sessions

INTERVENTIONS:
Behavioral: group cognitive behavioral therapy sessions — 12 group CBT sessions based on catching and challenging cognitive errors and behavioral techniques to deal with substance use problems
  Arms: CBT intervention arm

SUMMARY:
Aim of the study: In this study, the change in emotional intelligence will be assessed before and after group CBT sessions in male patients with substance use disorder in the inpatient department of the addiction unit at Mansoura University Hospital.

DETAILED DESCRIPTION:
Between the ages of fifteen and sixty-four, 5% of the global population, or nearly 200 million people, reported consuming at least one illegal substance per year. According to the 2008 World Drug Report, cannabis has a prevalence of 3.8%, compared to 0.6% for amphetamines and opiates, 0.3% for cocaine and heroin, and 0.2% for ecstasy. A cross-sectional study by [1] in Egypt with 2552 participants found that sedatives (8.7%) were the most commonly abused drugs, followed by alcohol (6.7%), cannabinoids (6.6%), and tramadol (2.4%). The prevalence of drug use was 8.9% for cigarette smoking followed by sedatives (4.3%), hashish (3.6%), alcohol (2.7%), cannabinoids (1.4%,) and tramadol (1.0%).

Lander et al. [2] believed that substance use disorder (SUD) is one of the most severe psychosocial traumas posing environmental, psychological, behavioral, and emotional challenges to individuals. It can cause obstacles for persons, families, and cultural foundations, endangering countries' dynamics. SUD is a brain disorder that impacts the person's behavior, manifests as psychological and physiological symptoms; and persists for a long duration despite its harmful and detrimental consequences.

Previous research has shown that different factors impact starting and following addiction. These factors are; 1) Individuals, such as the presence or lack of personality traits that make an individual vulnerable to addiction, for example, non-assertiveness as an individual factor. 2) Social factors, such as parental addiction, lack of parental control, availability of substances, presence of addicted peers, and so on [3].

Emotional intelligence (EQ) is a relatively recent behavioral model rising to prominence with Daniel Goleman's 1995 Book called 'Emotional Intelligence'. The early emotional intelligence theory was originally developed during the 1970s and 80s by the work and writings of psychologists Howard Gardner (Harvard), Peter Salovey (Yale), and John 'Jack' Mayer (New Hampshire) [4]. Emotional intelligence consists of the ability to motivate individuals such as endurance against frustration, impulse control, mood modification, and avoiding destructive stress to prevent mental disorders [5].

Emotional intelligence is a set of non-cognitive skills and abilities that can help a person deal with environmental stressors, according to [6]. Azzam and Elghonemy's [7] research demonstrated that emotional regulation was associated with mood improvement and a higher likelihood of SUD recovery. They found emotional intelligence to be an important factor in the treatment of substance use. [8] suggested that improvements in EI through treatment interventions can be an effective way to improve not only EI but also psychiatric symptoms both for the short term and the long term after rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with DSM5 diagnosis of substance use disorder
2. Age range 18 to 55 years
3. Agreeing to participate in the research and giving written informed consent
4. Average IQ as evidenced by the Wechsler Adult Intelligence scale

Exclusion Criteria:

1. Psychiatric comorbidities
2. Any neurological or medical conditions interfering with the cognitive abilities

4-Illiterate patients

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
emotional intelligence | 6 months
  Trait Emotional Intelligence Questionnaire (TEIQue-SF):
  The Trait Emotional Intelligence Scale (Petrides, 2009b) includes 30 items that assess the following four factors: well-being, self-control, sociability (each with six items), and emotionality (eight items), as well as four additional items 3, 14, 18, and 29, which do not belong to any factor and directly contribute to the evaluation of the overall degree of the trait emotional intelligence, as indicated by the scoring key. The questionnaire is graded on a seven-point Likert scale, with responses ranging from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating higher emotional intelligence. This TEIQue-SF scale has been used in numerous studies (Cooper & Petrides, 2010; Perera, 2015) owing to its good psychometric properties. The Arabic version was validated by Al-Dassean, (2023).

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction Unit, Psychiatry Department, Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Kabbash I, Zidan O, Saied S. Substance abuse among university students in Egypt: prevalence and correlates. East Mediterr Health J. 2022 Jan 31;28(1):31-40. doi: 10.26719/emhj.22.001. PMID 35165876
- [Background] Lander L, Howsare J, Byrne M. The impact of substance use disorders on families and children: from theory to practice. Soc Work Public Health. 2013;28(3-4):194-205. doi: 10.1080/19371918.2013.759005. PMID 23731414
- [Background] 3-Sho'aKazemi M. The comparative analysis of the relationship between coping strategies and attitude toward drug addicts (Persian). Addiction Studies; 2008.
- [Background] 4-Nazari K, Emami M. Emotional Intelligence: Understanding, applying, and measuring. Journal of Applied Sciences Research. 2012;8(3):1594-1607.
- [Background] 5-Bar-on R. The Emotional Quotient Inventory (EQ-i). A Test of Emotional Intelligence. Jossey. Bass; 2006.
- [Background] 6-Shareh, H., & Foshtanqi, K. (2019). The role of emotional intelligence and marital satisfaction in women's quality of life: Structural equation modeling. Journal of Fundamentals of Mental Health, 21(2), 109-120.
- [Background] 7-Azzam H, Elghonemy S. Emotional intelligence and substance abuse: A possible relation. Current Psychiatry. 2008; 15:113.25.
- [Background] 8-Henning, C., Crane, A. G., Taylor, R. N., & Parker, J. D. (2021). Emotional intelligence: relevance and implications for addiction. Current Addiction Reports, 8, 28-34.